CLINICAL TRIAL: NCT04277091
Title: The Effect of Upper-body High-intensity Interval Exercise vs. Moderate-intensity Continuous Exercise on Postprandial Metabolism
Brief Title: Upper-body High-intensity Interval Training and Mixed Meal Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Bilzon, Professor, University of Bath
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EP 18/19 087
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: High-Intensity Interval Training
Keywords: postprandial metabolism
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No exercise
- High-intensity interval exercise (Experimental): 10 x 60 s intervals at 80% peak power output (interspersed with 60 s recovery intervals at 10% peak power output)
  Interventions: Other: High-intensity interval training
- Moderate-intensity continous exercise (Experimental): 50% peak power output (duration determined to elicit same energy expenditure as high-intensity interval exercise condition)
  Interventions: Other: Moderate-intensity continuos training

INTERVENTIONS:
Other: High-intensity interval training — Arm-cranking exercise
  Arms: High-intensity interval exercise
Other: Moderate-intensity continuos training — Arm-cranking exercise
  Arms: Moderate-intensity continous exercise

SUMMARY:
Cycling and running-based high-intensity interval training are well-established to improve a variety of health outcomes. However, the efficacy of upper-body high-intensity interval training, vital for individuals with lower-body impairments, has yet to be well-characterized. The purpose of this study is to compare the effect of a single bout of upper-body high-intensity interval exercise (HIIE) in comparison to traditional moderate-intensity continuous exercise (MICE) on the blood response (e.g. glucose, insulin, fats) following a meal.

This study is recruiting able-bodied adults (aged 18-65 years). Participants will need to attend the laboratory at the University of Bath for two preliminary sessions, and three main study trials.

DETAILED DESCRIPTION:
The aim of this research is to determine the metabolic responses to a mixed-meal tolerance test following an acute bout of HIIE and an energy-matched MICE bout in able-bodied persons. The hypothesis is that HIIE and MICE will be more effective at reducing the total triglyceride responses compared to a resting control condition.

Preliminary measurements:

Preliminary testing will include measurements of weight and height. There will also be an assessment of resting metabolic rate and maximal exercise capacity. On a second visit, a HIIE familiarisation session will be performed to determine total energy expenditure of the session. All of the exercise protocols will take place on an arm crank ergometer at the University of Bath.

Main trial days:

Before all main trials, participants will be asked to refrain from performing any strenuous physical activity in the 48-h prior (i.e. day 0 and 1) and consuming alcohol/caffeine in the 24-h prior (i.e. day 1). On day 1, participants will be asked to record/replicate their diet using a weighed food-diary. Participants will be asked perform exercise (HIIE and MICE only) at 18:00 on day 1, having consumed no food (other than plain water) from 14:00. They will be given a standardised dinner to eat at 20:00, and asked to avoid the ingestion of any further food (other than plain water) for the rest of the evening.

On day 2 and upon arrival to the laboratory, a cannula will be inserted into a vein, and a baseline blood sample and expired air sample will be taken. The participant will then be asked to consume a smoothie, consisting of peanut butter, banana, coconut oil, sugar, and chocolate-flavoured whey protein powder. The meal should be consumed within 10 minutes and blood samples will be taken from the cannula at 15, 30, 45 60, and 90 minutes and then at every hour for 5 hours after consumption of the meal to monitor changes in metabolic markers. Expired gas samples will also be taken hourly and indirect calorimetry will be used to estimate relative fat and carbohydrate metabolism in response to the meal.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker
* No history of cardiovascular, metabolic, or neuromuscular disease

Exclusion Criteria:

* Individuals with a nut allergy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Postprandial triglyceride concentrations | 5 hours
  Postprandial triglyceride concentrations in serum samples

SECONDARY OUTCOMES:
Postprandial glucose concentrations | 5 hours
  Postprandial glucose concentrations in serum samples
Postprandial insulin concentrations | 5 hours
  Postprandial insulin concentrations in serum samples
Postprandial substrate oxidation | 5 hours
  Postprandial substrate oxidation determined by indirect calorimetry
Rating of Perceived Exertion | HIIE: End of Warm-Up, 8 min, 12 min, 16 min, 20 min, 24 min. MICE: 0, 20, 40, 60, 80, 100% through exercise session (exact time points dependent on exercise time for each participant)
  Global, central, and local rating of perceived exertion (6-20) during exercise
Heart Rate | HIIE: End of Warm-Up, 8 min, 12 min, 16 min, 20 min, 24 min. MICE: 0, 20, 40, 60, 80, 100% through exercise session (exact time points dependent on exercise time for each participant)
  Heart rate during exercise
Affect | HIIE: End of Warm-Up, 8 min, 12 min, 16 min, 20 min, 24 min. MICE: 0, 20, 40, 60, 80, 100% through exercise session (exact time points dependent on exercise time for each participant)
  Affect measured through the Feeling Scale (FS) during exercise. FS is a one item scale ranging from +5 ("Very good") to -5 ("Very bad").
Exercise Enjoyment | 30 min post-exercise
  Enjoyment measured by the Physical Activity Enjoyment Scale (PACES). PACES is a 17-item scale, with each item scored from 1 to 7. The total score will be calculated.
Self-efficacy | 30 min post-exercise
  Confidence in ability to perform exercise performed during trial in the next 4 weeks measured using a 5-item scale ranging from 0% ("Not at all" to 100% ("Extremely confident").

CONTACTS AND LOCATIONS:
Overall Officials: James Bilzon, Principal Investigator — University of Bath
Locations (1):
- Department for Health, Bath, United Kingdom